CLINICAL TRIAL: NCT00590330
Title: Microbial Community Composition and Dynamics in Lungs of Cystic Fibrosis Sibling Pairs
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Thomas Martin, MD, Children's Hospital, Boston
Other Study IDs: X07-10-0407
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — sputum or throat culture
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify all the bacterial species present in the respiratory tracts of patients with Cystic Fibrosis (CF), and to connect them with clinical information. Traditional culture methods of throat swab and sputum samples can only identify the most prevalent bacteria in samples, those of which there are over about 5 million bacteria per teaspoon. A recently developed method has been found to be more sensitive and can detect up to several hundred bacterial species in throat swab or sputum sample of individual CF patients.

DETAILED DESCRIPTION:
This study does not include testing of any investigational drugs and this is a noninvasive study requiring only a sputum/swab sample paired with information contained in the routine clinic letters and laboratory results your CF physicians obtain at your regular clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 1-16 upon enrollment
* Diagnosis of Cystic Fibrosis

Exclusion Criteria:

* None

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pulmonary clinic
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To identify all the bacterial species present in the respiratory tracts of patients with Cystic Fibrosis (CF). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Martin, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital, Boston, Massachusetts, United States